CLINICAL TRIAL: NCT05795595
Title: A Phase 1/2, Open-label, Multicenter, Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Anti-CD70 Allogeneic CRISPR-Cas9-Engineered T Cells (CTX131) in Adult Subjects With Relapsed or Refractory Solid Tumors
Brief Title: A Safety and Efficacy Study Evaluating CTX131 in Adult Subjects With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-005
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Clear Cell Renal Cell Carcinoma; Cervical Carcinoma; Esophageal Carcinoma; Pancreatic Adenocarcinoma; Malignant Pleural Mesothelioma
Keywords: CAR-T; Allogeneic; Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Uterine Cervical Neoplasms; Esophageal Neoplasms; Mesothelioma, Malignant; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX131 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX131

INTERVENTIONS:
Biological: CTX131 — CTX131 (CD70-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components)

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study evaluating the safety and efficacy of CTX131™ in subjects with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
An open-label, multi-center Phase 1/2 study of CTX131 in subjects with relapsed/refractory solid tumors. CTX131 is an is allogeneic CD70- directed chimeric antigen receptor (CAR) T cell immunotherapy comprised of allogeneic T cells that are genetically modified ex vivo using CRISPR-Cas9 (clustered regularly interspaced short palindromic repeats/ CRISPR associated protein 9) gene editing components (single guide RNA and Cas9 nuclease).

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years.
2. Unresectable or metastatic, relapsed/refractory, clear cell renal cell carcinoma, cervical carcinoma, pancreatic adenocarcinoma, esophageal carcinoma, and malignant pleural mesothelioma.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Adequate renal, liver, cardiac and pulmonary organ function.
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX131 infusion.

Key Exclusion Criteria:

1. Prior treatment with anti-CD70 targeting agents
2. History of certain central nervous system (CNS), cardiac or pulmonary conditions.
3. Presence of uncontrolled bacterial, viral, or fungal infection.
4. Active HIV, hepatitis B virus or hepatitis C virus infection.
5. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
6. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation): Incidence of adverse events | From CTX131 infusion up to 28 days post-infusion
  Defined as dose-limiting toxicities
Phase 2 (Cohort Expansion): Objective response rate (ORR) | From CTX131 infusion up to 60 months post-infusion
  ORR based on Independent Review Committee (IRC) assessment, defined as the proportion of subjects who have achieved a best overall response of CR or PR according to appropriate response evaluation criteria for each disease histology

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site 3, Duarte, California
  - Research Site 7, Chicago, Illinois
  - Research Site 6, Boston, Massachusetts
  - Research Site 2, St Louis, Missouri
  - Research Site 4, Durham, North Carolina
  - Research Site 1, Nashville, Tennessee
  - Research Site 5, Houston, Texas

IPD SHARING:
Plan to Share IPD: No